CLINICAL TRIAL: NCT00212537
Title: Disease Modifying Genes in Severe Asthma
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: H9698
Record Dates: First submitted 2005-09-19; First posted 2005-09-21 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Asthma
Keywords: Asthma and normal
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The total amount of blood drawn is approximately 5 tablespoons (75 ml). The blood sample will be processed to isolate "genetic material" (mainly DNA, RNA and protein). This genetic material will be used to try to identify the "genetic factors" or genes that a person inherits that make him or her more likely to develop asthma. The blood is used to test for allergies to weeds, trees, insects and molds (RAST) and a complete blood count.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gene and protein bank to study disease modifying and susceptibility genes and proteins in urban patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and above

Exclusion Criteria:

* Greater than 10 pack year tobacco history
* Lung diseases other than asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All individuals approached for participation in the Research Registry shall be able to read or comprehend English. Since participation in the Research Registry does not involve a risk of physical harm, women of childbearing potential will not be queried as to pregnancy status or tested for pregnancy unless they are requested to undergo a methacholine challenge test. There are no additional inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 941 (Actual)
Dates: Start 2002-04-08 (Actual); Primary Completion 2011-01-13 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
To recruit and characterize a cohort of subjects with asthma who reside in a high pollution, high asthma risk neighborhood | five yeARS

CONTACTS AND LOCATIONS:
Overall Officials: Joan Reibman, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Patrawalla P, Kazeros A, Rogers L, Shao Y, Liu M, Fernandez-Beros ME, Shang S, Reibman J. Application of the asthma phenotype algorithm from the Severe Asthma Research Program to an urban population. PLoS One. 2012;7(9):e44540. doi: 10.1371/journal.pone.0044540. Epub 2012 Sep 13. PMID 23028556
- [Derived] Liu M, Rogers L, Cheng Q, Shao Y, Fernandez-Beros ME, Hirschhorn JN, Lyon HN, Gajdos ZK, Vedantam S, Gregersen P, Seldin MF, Bleck B, Ramasamy A, Hartikainen AL, Jarvelin MR, Kuokkanen M, Laitinen T, Eriksson J, Lehtimaki T, Raitakari OT, Reibman J. Genetic variants of TSLP and asthma in an admixed urban population. PLoS One. 2011;6(9):e25099. doi: 10.1371/journal.pone.0025099. Epub 2011 Sep 22. PMID 21966427
- [Derived] Reibman J, Marmor M, Filner J, Fernandez-Beros ME, Rogers L, Perez-Perez GI, Blaser MJ. Asthma is inversely associated with Helicobacter pylori status in an urban population. PLoS One. 2008;3(12):e4060. doi: 10.1371/journal.pone.0004060. Epub 2008 Dec 29. PMID 19112508